CLINICAL TRIAL: NCT04795063
Title: Randomized Controlled Trials on Clinical Outcomes of Total Robotic Versus Robotic Assisted Distal Gastrectomy for Gastric Cancer
Brief Title: Total Robotic Versus Robotic Assisted Distal Gastrectomy for Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-022
Record Dates: First submitted 2021-03-04; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Gastric Cancer; Robotic Gastrectomy
Keywords: Gastric Cancer; robotic assisted distal gastrectomy; total robotic distal gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Robotic Distal Gastrectomy (Experimental): After exploration and randomization, patients received total robotic distal gastrectomy
  Interventions: Procedure: Total Robotic Distal Gastrectomy
- Robotic-Assisted Distal Gastrectomy (Active Comparator): After exploration and randomization, patients received robotic-assisted distal gastrectomy.
  Interventions: Procedure: Robotic-Assisted Distal Gastrectomy

INTERVENTIONS:
Procedure: Total Robotic Distal Gastrectomy — All the surgical procedures are performed using the robot system.
  Arms: Total Robotic Distal Gastrectomy
Procedure: Robotic-Assisted Distal Gastrectomy — After finishing the lymphadenectomy, the digestive tract reconstruction is performed extracorporal.
  Arms: Robotic-Assisted Distal Gastrectomy

SUMMARY:
To evaluate the clinical efficacy (safety, feasibility and long-term efficacy) of total robotic versus robotic assisted distal gastrectomy for patients with gastric cancer (cT1-4a, N0/+, M0).

DETAILED DESCRIPTION:
In the field of gastrectomy, Hashizume et al. first reported robotic gastrectomy in 2002. Since then, reports on the safety and feasibility of the application of robotic surgical system in the treatment of gastric cancer (GC) have gradually increased. Reports of robotic surgery for GC are increasing, especially in Asia. Several studies confirmed the advantages of robotic gastrectomy when compared with laparoscopic gastrectomy. However, whether total robotic gastrectomy is noninferior to robotic-assisted gastrectomy remains unclear. The investigator first carried out this study in the world to evaluate the efficacy of total robotic versus robotic assisted distal gastrectomy for GC.

ELIGIBILITY:
Inclusion Criteria:

1. Age from over 18 to under 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. cT1-4a (clinical stage tumor), N-/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
4. expected to perform distal gastrectomy with D1+/D2 lymph node dissection to obtain R0 resection surgicall results.
5. Performance status of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale
6. American Society of Anesthesiology (ASA) class I to III
7. Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
4. History of previous gastric surgery (except Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection (ESD/EMR) for gastric cancer)
5. Gastric multiple primary carcinoma
6. Enlarged or bulky regional lymph node （diameter over 3cm）supported by preoperative imaging
7. History of other malignant disease within the past 5 years
8. History of previous neoadjuvant chemotherapy or radiotherapy
9. History of unstable angina or myocardial infarction within the past 6 months
10. History of cerebrovascular accident within the past 6 months
11. History of continuous systematic administration of corticosteroids within 1 month
12. Requirement of simultaneous surgery for other disease
13. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
14. Forced expiratory volume in 1 second (FEV1)<50% of the predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity rates | 30 days
  This is for the early postoperative complication, which defined as the event observed within 30 days after surgery.

SECONDARY OUTCOMES:
3-year disease free survival rate | 36 months
  3-year disease free survival rate
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
overall postoperative serious morbidity rates | 30 days
  Refers to the incidence of early postoperative complication which is graded as Clavien-Dindo IIIA or higher
Total Number of Retrieved Lymph Nodes | 1 day
  Total Number of Retrieved Lymph Nodes
postoperative recovery course | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
postoperative nutritional status | 3, 6, 9 and 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status.
inflammatory immune response | Preoperative 3 days and postoperative 1, 3, and 5 days
  The variation of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response
Time of digestive tract reconstruction | 1 day
  From the beginning to the end of digestive tract reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Chang-ming Huang, MD, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China